CLINICAL TRIAL: NCT05632978
Title: An Observational Study of Epilepsy: Biology and Outcomes Using Real-world Data
Status: Recruiting | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Other Study IDs: 8345
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn more about phenotypic, genetic, biochemical, neurophysiological and radiological patterns in epilepsy.

Participants will be asked to consent to use of clinical and paraclinical data (obtained during standard care) for research, and will be asked to donate blood samples at their routine clinic visits.

DETAILED DESCRIPTION:
This is an observational study of people with epilepsy seen in South Wales, which will employ quantitative methods of analysis to meet the study aims. The study will build upon data already collected during routine clinical appointments from people with epilepsy who have come into contact with the National Health Service (NHS) epilepsy service at Cardiff & Vale University Health Board. The epilepsy service has clinical data on over 5000 people with epilepsy, and biological samples on approximately 400 people through the Welsh Neuroscience Research Tissue Bank.

The investigators propose to approach individuals being seen in the epilepsy clinics to gain consent for access to their routinely collected clinical and paraclinical data, and prospective donation of biological samples (predominantly blood samples, though consent will be sought for surplus brain tissue and cerebrospinal fluid (CSF) if brain surgery or lumbar puncture are being performed as part of clinical care, as well as hair, nail, and urine in some circumstances). This will enable a comprehensive disease register of a population-based sample of people with epilepsy to be established.

Interrogating the clinical and paraclinical data will allow investigation into clinical phenotypes, short- and long-term outcomes in epilepsy, and the relationship of clinical, demographic and biological variables. Biological samples will allow biochemical and genetic analysis of potential markers of disease, clinical phenotype, and prediction of outcomes including treatment responses, and allow contribution to the Epi25 international collaborative (http://epi-25.org/).

Inclusion in the study will involve no change to the normal clinical care or treatment of participants (except where participants choose to provide biological samples), and additional clinic visits will not be required outside of standard NHS care.

ELIGIBILITY:
Inclusion Criteria:

* Individual is being investigated for epilepsy and under the clinical care of the epilepsy unit at Cardiff & Vale University Health Board or regional clinics in Cwm Taf.
* Individual is at least 16 years old.
* Informed consent sought and given by individual.

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All people over 16 years old being investigated or followed-up for epilepsy.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Establish population-based cohort of people with epilepsy | 10-years
  Establish a population-based cohort of people with epilepsy and associated real-world clinical, paraclinical and biological data.

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Hamandi, Principal Investigator — Cardiff & Vale University Health Board
Locations (1):
- Cardiff and Vale UHB, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No